CLINICAL TRIAL: NCT00177788
Title: Voriconazole as Prophylaxis for Liver Transplant Recipients
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB # 0508150
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2012-08

CONDITIONS: Fungemia; Mycoses
Keywords: liver transplant; voriconazole prophylaxis; liver transplantation; voriconazole
MeSH Terms: conditions — Fungemia; Mycoses

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The study aims to determine if voriconazole prevents invasive fungal infections in liver transplant recipients. Endpoints would be: occurrence of invasive fungal infection and fungal colonization. Two groups will be compared: patients who received voriconazole as prophylaxis and historical controls who did not receive this prophylaxis.

DETAILED DESCRIPTION:
The following variables will be followed: time and location of positive cultures, underlying diseases and severity of illness, voriconazole usage prophylactically, physical exam findings, laboratory and radiographical data, antimicrobial usage, microbiological data and resistance patterns, choice of antifungal drugs once organism identified, suspected source of infection, microbiological outcomes, laboratory results, demographic information, medications, clinical outcome, gender, weight, ethnicity, and past medical history.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving a liver transplant at University of Pittsburgh Medical Center (UPMC) between January 1, 2001 and June 30, 2005.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: liver transplant patients receiving voriconazole
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2005-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Paterson, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States